CLINICAL TRIAL: NCT05996419
Title: Improving Psychosocial Functioning Among Veterans With Social Anxiety: A Pilot Evaluation of Self-Monitoring Intervention to Reduce Safety Behaviors
Brief Title: Intervention to Reduce Safety Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Ralph H. Johnson VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D4401-P; 121RX004401-01-A1 (Other Grant/Funding Number: Department of Veterans Affairs)
Record Dates: First submitted 2023-08-09; First posted 2023-08-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Social Anxiety
Keywords: Veteran; Social Anxiety; workforce

STUDY DESIGN:
Intervention Model Description: open trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DSB-Intervention (Experimental): Active intervention group receives text message intervention via ANNIE for 30 days
  Interventions: Other: DSB-I

INTERVENTIONS:
Other: DSB-I — Participant will receive text message every other day during active phase (30days) via ANNIE text messaging app related to the safety behaviors they identified prior to start.

SUMMARY:
Social anxiety is associated with significant deficits in social and occupational functioning. The proposed study seeks to evaluate the feasibility of implementing a brief text-based intervention for decreasing social anxiety related safety behaviors among Veterans attempting to re-integrate into the workforce. Findings from this pilot will support a larger randomized controlled study examining the efficacy of the intervention for improving functional outcomes and quality of life among Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Active enrollment in Compensated Work Therapy
* Score of > 25 on the Social Phobia Inventory
* Score of > 47 on the Subtle Avoidance Frequency Examination

Exclusion Criteria:

* Concurrent enrollment in another study related to social anxiety or improving functional status
* Recent (<3 month) history of psychiatric hospitalization, detoxification admission, or suicide attempt

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Subtle Avoidance Frequency Examination (SAFE) | Baseline and immediately after intervention
  32-item self-report measure designed to assess the frequency of safety behavior (SB) use. Respondents are asked to rate how often they engage in SBs such as "Rehearse sentences in your mind" and "Avoid eye contact" on a scale of 0 (Never) to 4 (Always). Scores on the SAFE range from 0-128 with higher scores indicative or more safety behavior use. total mean score
Social Phobia Inventory (SPIN) | baseline and immediately after intervention
  17-item measure of social anxiety severity. Participants are asked to rate items such as "I avoid doing things or speaking to people for fear of embarrassment" on a Likert-type scale of 0 (Not at all) to 4 (Extremely). Scores on the SPIN range from 0 to 68 with higher scores indicative of more severe social anxiety, total mean score

OTHER OUTCOMES:
General Self-Efficacy Scale (GSE) | Baseline and immediately after intervention
  10-item self-report measure of self-efficacy. The GSE demonstrates adequate internal reliability and convergent and divergent validity. Items range from 1 to 4 with total scores ranging between 10 and 40 and higher scores indicative of more self-efficacy;, total mean score
PTSD Checklist (PCL-5) | Baseline and immediately after intervention
  20-item instrument that parallels DSM-5 criteria for PTSD. Each item has five response options. Scores range from 0-80 with higher scores indicative of PTSD. Measures DSM-5 criteria for PTSD
Patient Health Questionnaire (PHQ-9) | Baseline and immediately after intervention
  a brief questionnaire that scores each of the 9 DSM-IV criteria for depression as "0" (not at all) to "3" (nearly every day). PHQ-9 score > or =10 have a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe, and severe depression, respectively , total mean score
Quality of Life Scale (QOL) | Baseline and immediately after intervention
  16-item self-report measure of quality of life across 5 conceptual domains: material and physical well-being, relationships with other people, social/community activities, personal development and fulfillment, and recreation, as well as an item on independence. The QOL demonstrates strong internal reliability and validity across medical populations and settings
Rate of recruitment | 18 month (end of recruitment)
  Proportion of veterans who agree to participate compared to total number approached for enrollment
THE VETERANS RAND 12-ITEM HEALTH SURVEY (SF-12) | Baseline and immediately after intervention
  valid and reliable instrument to measure quality of life/functional status in Veterans
Rate of retention | 18 month (end of recruitment)
  Number of veterans who enroll and complete study procedures as well as follow up interview compared to number who enroll
Credibility and Expectancy Questionnaire (CEQ) | Baseline
  will be used to assess the perceived credibility and expectancy related to effectiveness of the intervention. The CEQ will be administered only at baseline (following the intervention description), and 3 items from the measure will be used. These include: 1) how logical the program seems; 2) how successful the Veteran believes the program will be for him or her; and 3) how confident the Veteran would be recommending the program to a friend with similar needs.
Reactions to the Intervention | immediately after intervention
  This form consists of 3 questions comparable in scaling (i.e., using a 1 to 9 scale) to the CEQ. Specific questions target 1) satisfaction with the program; 2) likelihood of recommending the program to someone else; and 3) degree to which the Veteran believes the program helped with his or her difficulties and/or goals.

CONTACTS AND LOCATIONS:
Overall Officials: Anouk L. Grubaugh, PhD MA BS, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No